CLINICAL TRIAL: NCT04000607
Title: Exploratory Study of the Edwards APTURE Transcatheter Shunt System (ALT-FLOW Canada)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-11
Record Dates: First submitted 2019-06-24; First posted 2019-06-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Edwards APTURE transcatheter shunt system (Experimental)
  Interventions: Device: APTURE transcatheter shunt

INTERVENTIONS:
Device: APTURE transcatheter shunt — Transcatheter treatment of symptomatic left heart failure patients

SUMMARY:
The Exploratory study of the Edwards APTURE transcatheter shunt system (APTURE system) is a multi-center, prospective, exploratory study to evaluate initial clinical safety, device functionality, and effectiveness of the APTURE system.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic HF:

  * NYHA II w/ history of > II; III; or ambulatory IV AND
  * ≥1 HF hospitalization OR treatment with IV or oral diuresis within 12 months OR Elevated NT-proBNP value > 150 pg/ml in normal sinus rhythm, >450 pg/ml in atrial fibrillation, OR a BNP value > 50 pg/ml in normal sinus rhythm, > 150 pg/ml in atrial fibrillation within the past 6 months prior to study entry
* On stable GDMT for HF
* Left Ventricular Ejection Fraction (LVEF) ≤ 40% as determined by site cardiologist
* Hemodynamic criteria

  o At rest: Elevated LAP (or PCWP) > 15 mmHg AND LAP > RAP + 5 mmHg AND/OR supine ergometer exercise: elevated LAP (or PCWP) > 25 mmHg AND LAP > RAP + 10 mmHg
* Pulmonary Vascular Resistance (PVR) < 5.0 WU as determined by site cardiologist

Exclusion Criteria

* Severe HF:

  * NYHA IV, stage D, non-ambulatory, transplant list
  * Cardiac index ≤ 1.5 L/min/m2
  * Left Ventricular End-Diastolic Diameter (LVEDD) > 8 cm
  * LVEF <20%
* Valve disease

  * MR >3+ or > moderate MS, TR >3+ (severe on 5-point scale), AR >2+,
  * OR > moderate AS
* MI or therapeutic invasive cardiac procedure < 3 months
* TIA, stroke, CRT implanted < 6 months
* RV dysfunction > mild by TTE OR TAPSE <1.2 OR RV size ≥ LV size by TTE, OR Right Ventricular Fractional Area Change (RVFAC) ≤ 25%
* Dialysis OR renal dysfunction (S-Cr > 220 micromol/L OR e-GFR < 25ml/min/1.73 m2)
* 6MWT <50m OR >400m
* Active endocarditis or infection < 3 months
* Mean Right Atrial Pressure (mRAP) > 15 mmHg as determined by site cardiologist
* Body Mass Index (BMI) ≥ 45 kg/m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2019-07-10 (Actual); Primary Completion 2023-11-03 (Actual); Study Completion 2028-11-11 (Estimated)

PRIMARY OUTCOMES:
Rate of major cardiac/cerebrovascular/renal events and re-intervention (Safety Endpoint) | 30 Days
  Composite of major adverse cardiac, cerebrovascular, renal events (MACCRE) and re-intervention for study device related complications at 30 days.

SECONDARY OUTCOMES:
Rate at which device is successfully implanted (Device Success) | Day 0
  Device is deployed as intended and the delivery system is successfully removed as intended at the time of the patient's exit from the implant procedure room.
Rate at which device is patent and subject is discharged from hospital without the need for additional intervention for the device (Procedural Success) | 10 Days post-op
  Device success with evidence of shunt patency and hospital discharge without the need for additional surgical or percutaneous intervention related to the study device including unacceptable Qp/Qs values.
Rate at which the procedure is successful without major cardiac/cerebrovascular/renal events and re-intervention (Clinical Success) | 30 Days
  Procedural success without major adverse cardiac, cerebrovascular, and renal events (MACCRE) and re-intervention for study device related complications at 30 days.
Change in the ratio of systemic blood flow (Qs) to the pulmonary blood flow (Qp), called "Qp/Qs", from Baseline to Follow Up | 3 Months, 6 Months
  Change in Qp/Qs value from Baseline to Follow Up (3Month, 6Month)
Change in pulmonary capillary wedge pressure (PCWP) from Baseline to Follow Up | 3 Months, 6 Months
  Change in PCWP value from Baseline to Follow Up (3Month, 6Month)
Change in mean systolic & diastolic pulmonary artery pressure (PAP) and change in mean right atrial pressure (RAP) from Baseline to Follow Up | 3 Months, 6 Months
  Change in PAP and RAP values from Baseline to Follow Up (3Month, 6Month) under the same test conditions (e.g. comparison in the value at rest at baseline, to at rest at follow up; comparison in the value at exercise at baseline, to at exercise at follow up)
Change in Pulmonary Vascular Resistance (PVR) from Baseline to Follow Up | 3 Months, 6 Months
  Change in PVR value from Baseline to Follow Up (3Month, 6Month) under the same test conditions (e.g. comparison in the value at rest at baseline, to at rest at follow up; comparison in the value at exercise at baseline, to at exercise at follow up)
Change in two parameters related to Tricuspid Annular Plane Excursion (TAPSE) from Baseline to Follow Up | 3 Months, 6 Months
  Change in two parameters from Baseline to Follow Up (3Month, 6Month):
  1. "TAPSE", Tricuspid Annular Plane Excursion
  2. "TAPSE/sPAP", Tricuspid Annular Plane Excursion (TAPSE) divided by the systolic pulmonary Artery Pressure (sPAP)

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - St. Michael's Hospital, Toronto, Ontario